CLINICAL TRIAL: NCT05033470
Title: A Multicentre Prospective Study Evaluating an Off-loading Mattress Overlay System in Healing of Stage 3 Pressure Ulcers (DABIRPrU)
Brief Title: A Multicentre Prospective Study Evaluating an Off-loading Mattress Overlay System in Healing of Stage 3 Pressure Ulcers
Acronym: DABIRPrU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Dabir Surfaces Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DABITPrU-001
Record Dates: First submitted 2021-08-13; First posted 2021-09-02 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Multi-center prospective pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabir Surface Mattress Overlay System (Experimental): Eligible patients are treated with a mattress overlay system and standard of care (debridement, proper moisture balance, reduction of bacterial burden and nutritional counseling). Subjects will be seen weekly for 4 weeks. Patients who respond to the offloading device, may use the overlay for an additional 12 weeks with monthly follow-up visits in the clinic or their home. Subjects undergo study procedures on a weekly basis.
  Interventions: Device: Dabir Mattress Overlay System

INTERVENTIONS:
Device: Dabir Mattress Overlay System — Dabir Surface mattress overlay system consists of a controller and a low-profile alternating pressure (AP) surface (placed over a non-powered mattress) with hundreds of air-filled geometric nodes arranged in rows. . The multiple rows of nodes inflate and deflate in alternating sequence every five minutes. During deflation phase, the skin and soft tissues experience reduced pressure/loading and enhanced perfusion. In conjunction with Standard of Care: Debridement, Proper moisture balance, off-loading, reduce bacterial burden and nutritional counseling.
  Other Names: standard of care

SUMMARY:
This study will evaluate the use of a mattress overlay system to promote the healing of full thickness pressure ulcers. The overlay is placed over the patient's bed making it easier for patients to get in and out of bed. In addition, the overlay has blue tooth capabilities that will allow clinicians to remotely monitor adherence with the device.

DETAILED DESCRIPTION:
The study is a multi-center, prospective, study designed to evaluate the use of an alternating mattress overlay in the treatment of stage 3 pressure ulcers. After screening, eligible subjects will receive a mattress overlay system for the 4 weeks of treatment. The mattress is fitted to the patient's bed/mattress in his/her home or skilled nursing facility (SNF). Patients responding to the offloading regimen (percent wound area reduction >20% at 4 weeks) may use the overlay for up to 12 additional weeks. The SOC in this study is debridement, proper moisture balance, reduction of bacterial burden and nutritional counseling.

ELIGIBILITY:
Inclusion Criteria

1. Subjects are male or female, 18 years of age or older.
2. Pressure ulcer/injury present for greater than 4 weeks (documented in the medical record).
3. Subject has clinical documentation of no visible wound improvement in the post four weeks of standard of care. Objectively, less than 20% healing in the past four weeks from the first treatment visit.
4. Study ulcer is a minimum of 2.0 cm2 and a maximum of 50 cm2 at first treatment visit.
5. The subject is able and willing to follow the protocol requirements.
6. Subject has signed informed consent.

Exclusion Criteria

1. Subject has major uncontrolled medical disorder such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.
2. Subject currently being treated for an active malignant disease or subjects with history of malignancy within the wound.
3. The Subject has other concurrent conditions that, in the opinion of the Investigator, may compromise subject safety.
4. Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
5. Subject is pregnant or breast feeding.
6. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
7. Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the l 30 days preceding the first treatment visit.
8. Affected extremity requiring hyperbaric oxygen during the trial or within 2 weeks of treatment visit 1.
9. Known HbA1C >12%.
10. Mini-nutritional assessment Malnutrition Indication score <17.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Wound Reduction in Surface Area | 4 week
  The percentage change in ulcer size (wound area reduction) from baseline to 4 week completion

SECONDARY OUTCOMES:
Pain assessment | 4 weeks
  Assessment of the pain level linked to the wound, using a numeric pain scale. Numeric Pain Scale from 0-10 anchored by word descriptors at each end. A numerical scale will be used to assess pain. Subject will be asked to indicate a numerical value that best represents the pain intensity at ulcer site on a scale of 0 to 10 anchored by "word descriptors" at each end, as "no pain" on the left side and "worst possible pain" on the right side of the number line. The number 0 represents "no pain", the number 5 represents "moderate pain" and the number 10 represents the "worst possible pain". The subject indicates the level of pain intensity by selecting a number on the line that represents their perception of their current state.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Serena, Study Director — cro
Locations (1):
- SunnyView, Butler, Pennsylvania, United States